CLINICAL TRIAL: NCT05736471
Title: Computational Dissociation of the Causes of Cognitive Rigidity in Depression
Brief Title: Cognitive and Affective Processes Online
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: Psych-2020-28403
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Depression
Keywords: Cognitive rigidity; Foraging; Exploration-Exploitation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test Group: involves a single testing session with surveys and tasks relevant to the experiment involving behavioral tasks and self-report questions through an online crowd-sourcing platform
  Interventions: Diagnostic Test: Computational dissociation of the causes of cognitive rigidity in depression

INTERVENTIONS:
Diagnostic Test: Computational dissociation of the causes of cognitive rigidity in depression — involves a single testing session with surveys and tasks relevant to the experiment involving behavioral tasks and self-report questions through an online crowd-sourcing platform

SUMMARY:
This study will provide data for evaluating the psychometric characteristics of the tests assessing cognitive flexibility, including their (1) internal consistency, (2) feasibility and tolerability, their (3) convergent and discriminant validity of cognitive and affective constructs such as those introduced to understand mental disorders, and (4) sensitivity (and correspondence) to individual differences. For these tests to be useful in studying clinical conditions, they must show adequate reliability, validity, and sensitivity in large samples of convenience.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* English-speaking
* Live in the U.S.
* Have access to an internet connected computer
* Users of the mTurk and Prolific survey website

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prolific online
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Relationship of cognitive rigidity to depressive symptoms | 1 hour
  Relationship of model-based measures of learning from the past and anticipating the future to symptoms of depression, specifically anhedonia
Relationship between environmental volatility and cognitive rigidity | 1 hour
  Relationship between environmental volatility and model-based measures of cognitive rigidity.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Herman, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States